CLINICAL TRIAL: NCT01476033
Title: Impact of Encapsulated Fruit, Berry and Vegetable Juice Powder Concentrate on Oxidative Stress, Inflammation and Blood Flow Before and Post Exercise in Overweight, Middle-aged, Women.
Brief Title: Strong Women Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Green Beat (Other)
Responsible Party: Principal Investigator, Lamprecht Manfred PhD, PhD, Principal investigator, Green Beat
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 23-508 ex 10/11
Record Dates: First submitted 2011-11-16; First posted 2011-11-22 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Oxidative Stress; Inflammation
Keywords: Oxidative stress; inflammation; blood flow
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fruit, berry and vegetable concentrate (Active Comparator): 20 ladies receive an encapsulated, powdered fruit, berry and vegetable concentrate for 8 weeks
  Interventions: Dietary Supplement: nutraceutical group
- 20 women with placebo (Placebo Comparator): placebo for 8 weeks
  Interventions: Dietary Supplement: nutraceutical group

INTERVENTIONS:
Dietary Supplement: nutraceutical group — 6 capsules of supplement or placebo for 8wk

SUMMARY:
The investigators investigate the impact of an encapsulated fruit, berry and vegetable juice powder concentrate on oxidative stress, inflammation and blood flow before and post exercise in overweight, middle-aged, women.

Main hypotheses (H1):

* The nutraceutical has an impact on oxidative stress reduction.
* The nutraceutical has an impact on inflammation.
* The nutraceutical has an impact on blood flow and microcirculation.
* Walking exercise for 30 minutes has an impact on oxidative stress- and inflammation markers.
* Walking exercise for 30 minutes has an impact on blood flow and microcirculation
* The combination of nutraceutical supplementation + walking exercise for 30 minutes has an impact on oxidative stress- and inflammation markers, and on blood flow/microcirculation.

ELIGIBILITY:
Inclusion Criteria:

* women
* BMI > 27
* praemenopausal
* non smokers
* eligibility for exercise
* 4wk wash out

Exclusion Criteria:

* male
* all people not matching this age group
* BMI > 40 and < 27
* peri- or postmenopausal women
* smokers
* all women taking dietary supplements
* all women that fail in ergometric exercise eligibility testing, refering to the standards in sports medicine (e.g.: significant ST-decrease or increase, blood pressure > 240 mmHg, tachycardia, polymorphic extrasystolia, cyanosis, bradyarrhythmia..)
* Diabetics
* osteoporosis or osteopenia

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Carbonyl groups on protein, oxidized LDL, Malondialdehyde, TNF-alpha, IL-6, Trombelastometry and peripheral microcirculation | 6 months
  Carbonyl groups on protein as indicators of protein oxidation; oxidized LDL, Malondialdehyde as indicators of Lipidoxidation; TNF-alpha, IL-6 as indicators of inflammation; Trombelastometry: clotting time, thrombocyte ahesion, trombocyte aggregation from whole blood as indicators for blood flow and hemostasis; Peripheral microcirculation in subcutis as indicator for blood flow in peripheral subcutis.

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Lamprecht, PhD PhD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria